CLINICAL TRIAL: NCT02413866
Title: Weight Outlooks by Restriction of Diet and Sleep
Acronym: WORDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Xuewen Wang, Assistant Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00036519
Record Dates: First submitted 2015-04-07; First posted 2015-04-10 (Estimated); Last update posted 2019-04-19 (Actual); Status verified 2016-12

CONDITIONS: Weight
Keywords: body composition; anthropometry
MeSH Terms: conditions — Body Weight | interventions — Sleep

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Calorie Restriction Only (Experimental): Participants in this group will be decreasing their caloric intake to approximately 95% of their resting metabolic rate. We will provide one meal for 4 days of the week, and participants will be required to keep an accurate dietary record of all food and drink. Participants assigned to this group will be instructed to keep a fixed sleep schedule based on their own sleep/napping habits.
  Interventions: Behavioral: Calorie restriction only
- Sleep & Calorie Restriction (Experimental): Participants in this group will decrease their caloric intake to approximately 95% of their resting metabolic rate in addition to reducing their total time in bed by 90 minutes 5 days a week.
  Interventions: Behavioral: Sleep & calorie restriction

INTERVENTIONS:
Behavioral: Calorie restriction only — Participants randomly assigned to this group will be instructed to reduce their daily energy intake to 95% of their resting metabolic rate.
  Arms: Calorie Restriction Only
Behavioral: Sleep & calorie restriction — Participants randomly assigned to this group will be instructed to reduce their total time in bed by 90 minutes 5 days a week, in addition to restricting their dietary intake to approximately 95% of their resting metabolic rate.
  Arms: Sleep & Calorie Restriction

SUMMARY:
The purpose of this study is to examine whether chronic moderate sleep restriction effects the amount of body fat and lean mass loss, and calorie expenditure, in individuals who are participating in a dietary weight loss program.

DETAILED DESCRIPTION:
Participants will be randomly assigned to an 8-week program of either restricted diet alone, or restricted diet with restricted sleep for 5 days a week. The total expected duration of participation is approximately 3 months.

ELIGIBILITY:
Inclusion Criteria:

* age between 35-55 years,
* BMI between 30-35 kg/meters squared,
* total sleep time between 6.5-8 hours

Exclusion Criteria:

* work requiring changing schedule,
* use of sleep aids or sleep medication

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2015-01; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
body composition measured via DXA scans | 4 months
  Body composition will be measured via DXA scans prior to intervention and post intervention to compare losses in lean body mass and fat mass.

CONTACTS AND LOCATIONS:
Overall Officials: Xuewen Wang, PhD, Principal Investigator — University of South Carolina
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

REFERENCES:
- [Derived] Sparks JR, Porter RR, Youngstedt SD, Bowyer KP, Durstine JL, Wang X. Effects of moderate sleep restriction during 8-week calorie restriction on lipoprotein particles and glucose metabolism. Sleep Adv. 2021 Jan 28;1(1):zpab001. doi: 10.1093/sleepadvances/zpab001. eCollection 2020. PMID 33644759
- [Derived] Wang X, Sparks JR, Bowyer KP, Youngstedt SD. Influence of sleep restriction on weight loss outcomes associated with caloric restriction. Sleep. 2018 May 1;41(5):10.1093/sleep/zsy027. doi: 10.1093/sleep/zsy027. PMID 29438540